CLINICAL TRIAL: NCT01259037
Title: A Study of Ultrasonography With Elastography in Skin Neoplasms
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Darius Mehregan, Chairman of Dermatology, Wayne State University
Other Study IDs: Elastography1
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Benign and Malignant Skin Neoplasms
Keywords: Elastography; Cutaneous; Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsies of lesions imaged with ultrasound are processed for routine histology and retained.

SUMMARY:
This study will look at high frequency ultrasound as a medical imaging modality and apply it to skin lesions. Elastography is an ultrasonic method of looking at the hardness of an area. We will use this to try and differentiate between benign and cancerous skin lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with skin lesions undergoing biopsy for diagnosis.

Exclusion Criteria:

* Patients with skin lesions which do not require biopsy for diagnosis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General dermatologic population from suburban referral clinic.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06-30 (Actual); Study Completion 2017-10-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States